CLINICAL TRIAL: NCT04367571
Title: The Effects of Osteopathic Manipulative Treatments on Neurogenic Bowel Dysfunction in Patients With Spinal Cord Injuries: a Randomized Manual Placebo Controlled Trial
Brief Title: Osteopathic Manipulative Treatments and Neurogenic Bowel Dysfunction in Patients With Spinal Cord Injuries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, head of rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSLCE/800/OMT
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental)
  Interventions: Other: Osteopathic Manipulative treatment (OMT)
- Manual Placebo (Placebo Comparator)
  Interventions: Other: Manual Placebo (MP)

INTERVENTIONS:
Other: Osteopathic Manipulative treatment (OMT) — OMT techniques were focused on correcting the dysfunctions found before each OMT session and included myofascial techniques, balanced ligamentous tension, visceral manipulations and osteopathy in the cranial field.
  OMT group will receive a total of 4 sessions, one time each week for 4 weeks. Each session will last 40 minutes. It will be required by the patients to modify their bowels habits. The subjects will be evaluated right at baseline (T0), after one month (T1) after four sessions (T2) and after 1 month after the treatment (T3).
  Arms: Osteopathic Manipulative Treatment
Other: Manual Placebo (MP) — The MP treatment consists of passive touch without joint mobilization in a protocolled order. The practictioners will be standing next to the bed, they'll touch lumbar and dorsal spine of the subjects in prone position for 10 minutes, and then in supine position, they'll touch for 10 minutes the shoulders, the hips, then the neck, the sternum and the chest for 5 minutes each.
  MP group will receive a total of 4 sessions, one time each week for 4 weeks. Each session will last 40 minutes. It will be required by the patients to modify their bowels habits. The subjects will be evaluated right at baseline (T0), after one month (T1) after four sessions (T2) and after 1 month after the treatment (T3).
  Arms: Manual Placebo

SUMMARY:
Studies based on the relationship between Osteopathic Manipulative Treatment (OMT) and the gastrointestinal system have been conducted in patients with constipation with Irritable Bowel Syndrome (IBS), and in children with infantile cerebral palsy. For IBS patients, OMT can facilitate visceral vascularization and restore the physiological elasticity and motility of the viscera, and of the peritoneal structures around the viscera. The study also focused on the effects of OMT on women and constipated children, indicating an improvement in the stool consistency, reduction in the symptoms of constipation, the severity of the constipation, and in the use of laxative drugs.

In patients with Spinal Cord Injury (SCI), the secondary health disorders include the alteration of gastric acid secretion, abnormal colonic myenteric activity, and neurogenic bowel dysfunction (NBD). Patients with NBD present loss or absence of normal bowel function. About 80% of SCI is accompanied by NBD resulting in a lower quality of life caused by loss of independence, sense of embarrassment, mental disorder, social isolation.

Conservative treatments for NBD after SCI include oral laxatives, enemas, retroanal trans-grade irrigation and digital anorectal stimulation. These treatments are mainly focused on promoting intestinal faecal evacuation and on strengthening the anal sphincter to improve bowel function. There are no studies that investigate the effects of OMT on patients with SCI, however, several studies have already showed the effects of OMT on the nervous system, on the hemodynamic system, and on visceral motility. Therefore, the starting hypothesis of this study is to use OMT in order to improve the symptoms of NBD in subjects with SCI, through a global OMT

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old,
* chronic spinal cord injury (more than six months between the spinal injury and the enrollment in the research),
* injury classified per the ASIA impairment scale AIS A, B, C or D localized at a cervical-dorsal level up to D10.

Exclusion Criteria:

* Use of bowel emptying techniques such as retrograde trans-anal irrigation
* presence of previous inflammatory intestinal diseases
* metabolic or endocrinological dysfunctions,
* pregnancy state
* cognitive disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Neurogenic Bowel Dysfunction (NBD) | at 3 months
  NBD score changes from baseline at 3 moths. self-reported questionnaire. The Neurogenic Bowel Dysfunction is a 10-item questionnaire covering frequency of bowel movements, headache, perspiration or discomfort during defaecation; medication for constipation or faecal incontinence; time spent on defaecation; frequency of digital stimulation or evacuation; frequency of faecal incontinence; flatus; and perianal skin problems. It ranges between 0 and 47; lower scores indicate a better bowel function, while a score over 14 is considered to be an index of severe bowel dysfunction.
  Score 0-6 Very low 7-9 Low 10-13 Moderate 14 or more Severe The hypothesis of treatment efficacy is supported by the observation of a difference between the groups in the NBD score.

SECONDARY OUTCOMES:
Knowles Eccersley Scott Symptom (KESS) | at baseline, after one month, after 4 treatment sessions, one month after the last treatment
  KESS score changes from baseline at 3 months. The KESS is a validated questionnaire for diagnosis of constipation. KESS has an added advantage of differentiating between various subtypes of constipation. Total scores can range from 0 (no symptoms) to 39 (high symptom severity). A cut-off score of > 11 indicates constipation
Patient Assessment of Constipation Quality Of Life scale (PAC-QOL) | at baseline, after one month, after 4 treatment sessions, one month after the last treatment
  PAC-QOL score changes from baseline at 3 months. Each item of the 28-item questionnaire was scored on a 5-point Likert-type scale from 0 to 4, with (0 = none/not at all, 1 = a little bit/a little bit of the time, 2 = moderately/some of the time, 3 = quite a bit/most of the time, 4 = extremely/all the time). Scores were reported overall and for each of the four subscales (physical discomfort, psychosocial discomfort, worries and concerns, and satisfaction). An improvement (reduction) of ≥1 point in PAC-QOL score was considered clinically significant based on previous validation studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Lucia Foundation I.R.C.C.S., Roma, Rm, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Todd CL, Johnson EE, Stewart F, Wallace SA, Bryant A, Woodward S, Norton C. Conservative, physical and surgical interventions for managing faecal incontinence and constipation in adults with central neurological diseases. Cochrane Database Syst Rev. 2024 Oct 29;10(10):CD002115. doi: 10.1002/14651858.CD002115.pub6. PMID 39470206